CLINICAL TRIAL: NCT06826716
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study to Assess the Effect of Libifem® (VL-GF-01) on Fertility in Women With Diminished Ovarian Reserve
Brief Title: A Study to Assess the Effect of Libifem® (VL-GF-01) on Fertility in Women With Diminished Ovarian Reserve
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR/240801/IP/FF
Record Dates: First submitted 2024-12-17; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Female Fertility
MeSH Terms: interventions — fenugreek seed meal; maltodextrin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP(Trigonella foenum graecum)) (Experimental): Dose: 600 mg/day Regimen:
  One capsule (300 mg) to be taken twice a day 30 minutes post breakfast and dinner Route of administration: Oral
  Interventions: Dietary Supplement: Fenugreek (Trigonella foenum graecum)
- Placebo (Maltodextrin) (Placebo Comparator): Dose: 600 mg/day Regimen:
  One capsule (300 mg) to be taken twice a day 30 minutes post breakfast and dinner Route of administration: Oral
  Interventions: Dietary Supplement: Placebo (Maltodextrin)

INTERVENTIONS:
Dietary Supplement: Fenugreek (Trigonella foenum graecum) — Dose: 600 mg/day Regimen:
  One capsule (300 mg) to be taken twice a day 30 minutes post breakfast and dinner Route of administration: Oral
  Arms: IP(Trigonella foenum graecum))
Dietary Supplement: Placebo (Maltodextrin) — Dose: 600 mg/day Regimen:
  One capsule (300 mg) to be taken twice a day 30 minutes post breakfast and dinner Route of administration: Oral
  Arms: Placebo (Maltodextrin)

SUMMARY:
The present study is a randomized, double-blind, placebo-controlled, parallel clinical study. Approximately 156 participants will be screened, and considering a screening failure rate of 20%, not more than 124 participants will be randomized in a ratio of 1:1 to receive either Libifem® or placebo and will be assigned a unique randomization code. Each group will have not less than 50 completed participants after accounting for a dropout/withdrawal rate of 20%.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ready to give voluntary, written informed consent to participate in the study.
2. Women of age between 25 to 35 years who wish to conceive.
3. Women with BMI between 18.5 to 34.9 kg/m2 (both values included).
4. Women who are unable to conceive for at least one year with an unprotected sexual life.
5. Women engaging in sexual act regularly and agree to continue the same at least twice a week during the study.
6. Women with bilateral tubal patency as confirmed by reports (within last one year from screening) of Hysterosalpingography (HSG) or Sonosalpingography (SSG).
7. Eumenorrheic women with a regular menstrual cycle of 28 ± 5 days.
8. Women with Hemoglobin levels greater than or equal to 10 g/dL.
9. Women with Anti-Mullerian hormone (AMH) greater than 0 and less than 1.5 ng/ml on day 2 of menstrual cycle.
10. Females with serum Thyroid-stimulating hormone (TSH) levels between 0.4 mIU/L to 5 mIU/L [both values inclusive] with or without medication.
11. Women who are not pregnant during the time of screening as assessed by UPT.
12. Women who have never undergone IVF procedure.
13. Women with their male partners having an acceptable serum analysis report as per PI.
14. Women willing to complete all study-related assessments and to complete all clinical study visits as per the protocol.

Exclusion Criteria:

1. Any chronic illness like hyper-prolactinemia.
2. Females diagnosed with stage 3 and stage 4 Endometriosis.
3. Females with a history of recurrent pregnancy loss (defined as ≥ 2 failed clinical pregnancies before 22 weeks of gestational age).
4. Females clinically diagnosed with Polycystic Ovarian Syndrome (PCOS).
5. Females with a prior history (within the last 6 months from screening) of ≥3 cycles of ovulation induction.
6. History of ovarian hyper-response.
7. History of any endocrine abnormality (eg: Adrenal gland disorders, pituitary disorders, endocrine diseases, dyslipidemia, etc.).
8. Females previously diagnosed with hyperparathyroidism and/or hyperthyroidism.
9. Females with a history of any psychiatric disorder.
10. Currently undergoing or have previously undergone Hormone Therapy (HT) for treatment of fertility in the previous 6 months.
11. Currently consuming Ayurvedic/dietary supplements, and/or currently consuming steroids or if consumed in the last 3 months before screening.
12. Currently consuming cytotoxics and immunosuppressants.
13. History of uncontrolled hypertension and/or systolic blood pressure greater than equal to 140 mmHg and/or diastolic blood pressure greater than equal to 90 mmHg.
14. Fasting blood glucose (FBG) greater than or equal to 126 mg/dL.
15. Participation in other clinical studies in the past 3 months.
16. History of alcohol or drug abuse in the 12 months prior to screening.
17. History of cancer.
18. Hematological disorders.
19. History or presence of any Sexually Transmitted Disease (STD).
20. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential individual at risk because of participation in the study, or influences the results or the potential individual's ability to participate in the study.
21. History or presence of HIV, cardiovascular, gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e. Crohn's disease, short bowel, acute or chronic pancreatitis or pancreatic insufficiency).
22. Lactating women

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female fertility
Enrollment: 150 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of the Investigational product (IP) on time to pregnancy (TTP) as assessed by serum levels of Beta-human Chorionic Gonadotropin (Beta-hCG). | From Date of screening upto 6 month
  The mid-cycle surge in LH lasts 36-48 hours and triggers ovulation, which is the release of the egg from the follicle. The peak progesterone levels occur halfway through the last 14 days of the cycle, known as the luteal phase. Progesterone prepares the endometrium for potential implantation if the egg is fertilized and forms an embryo. If an embryo develops, it produces human chorionic gonadotropin (hCG), which activates the Luteinizing Hormone (LH) receptors and helps maintain the corpus luteum's function, allowing it to continue producing progesterone and supporting the pregnancy.
  When a participant misses her menstrual cycle after the expected cycle date, clinical pregnancy will be confirmed by the quantitative Beta-hCG test on the subsequent day 10 visi

SECONDARY OUTCOMES:
To assess the impact of the IP as compared to baseline and placebo on Ovulation status as assessed by Antral follicle count (AFC) using Transvaginal ultrasonography (TVS) (On day 2 & day 10 of each menstrual cycle) | From Date of screening upto 6 month
  The antral follicle count (AFC) evaluates the number of visible follicles in a woman's ovaries at the beginning of her menstrual cycle.The greater the number of visible follicles in the ovary, the higher the likely ovarian reserve. Women experiencing infertility are more likely to have lower antral follicle counts compared to those who are not infertile.TVS offers a precise and consistent measurement of the total number of antral follicles throughout the menstrual cycle.Thus, AFC will be assessed using TVS on days 2 and 10 of each menstrual cycle throughout the Study
To assess the impact of the IP as compared to baseline and placebo on Reduction in serum Follicle-Stimulating Hormone levels(On day 2 of each menstrual Cycle) | From Date of screening upto 6 month
  FSH levels are highest just before ovulation in the follicular phase and help in the development of the follicles. The levels decrease after the onset of menstruation because of the negative feedback mechanism of inhibin B and estrogen.
To assess the impact of the IP as compared to baseline and placebo on Reduction in serum Estradiol levels(On day 2 & day 10 of each menstrual cycle) | From Date of screening upto 6 month
  Like FSH, estradiol levels fluctuate throughout the menstrual cycle, reaching peaks in both the late follicular and mid-luteal phases. A reduction in the estradiol levels in the menstrual phase can lead to a replenished ovarian reserve. Thus, in the present study, the serum estradiol levels will be analyzed on day 2 and day 10 of each menstrual cycle throughout the study
To assess the impact of the IP as compared to baseline and placebo on Change in the ovarian reserve as assessed by serum Anti-Mullerian hormone levels [On day 2 of each menstrual cycle] | From Date of screening upto 6 month
  Anti-Mullerian Hormone (AMH). AMH is a sensitive biomarker of ovarian reserve, as its levels decline before FSH increases. This test demonstrates a strong correlation between the primordial follicle pool and ovarian response to stimulation .AMH has several advantages over traditional ovarian reserve markers: it is the first to change with age, shows minimal variability within a single cycle and between consecutive cycles, and can be measured at any point during the cycle.37 Therefore, in the present study, AMH levels will be analyzed on day 2 of each menstrual cycle throughout the study

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Sachi Hospital, Ahmedabad, Gujarat
  - Shardaben General Hospital, Ahmedabad, Gujarat
  - Imperial Multispeciality Hospital, Pune, Maharashtra
  - Ashwin Medical Foundations Moraya Multispeciality Hospita, Pune, Maharshtra
  - Jnu ,Jaipur, Jaipur, Rajashthan
  - Pragya Mother & Child care Hospital, Varanasi, Uttar Pradesh
  - Panchsheel Hospital Pvt. Ltd., Delhi

IPD SHARING:
Plan to Share IPD: No